CLINICAL TRIAL: NCT04624763
Title: Protection on Cardiac Function With Left Bundle Branch Pacing in Patients With Atrioventricular Block(OptimPacing)
Brief Title: Protection of Cardiac Function With Left Bundle Branch Pacing in Patients With Atrioventricular Block
Acronym: OptimPacing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: West China Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Shanghai Zhongshan Hospital (Other); Zhongshan Hospital Xiamen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Fujian Medical University Union Hospital (Other); Xijing Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Southwest Hospital, China (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FirstNanjingMU003
Record Dates: First submitted 2020-10-22; First posted 2020-11-12 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Atrioventricular Block
Keywords: Left bundle branch pacing; Atrioventricular block; Right ventricular pacing; Cardiac function
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBBP group (Experimental): In this arm, a left bundle branch pacing(LBBP) lead is attempted to be placed.
  Interventions: Procedure: Left bundle branch pacing
- RVP group (Active Comparator): In this arm, a right ventricular pacing(RVP) lead are placed.
  Interventions: Procedure: Right ventricular pacing

INTERVENTIONS:
Procedure: Left bundle branch pacing — LBBP is defined if fulfilling criterion 1 and at least one in criteria 2:
  1. Paced morphology of RBBD in surface lead V1 (QR, Qr, rSr', rSR' or Qrs);
  2. One of the following should be met:
     1. Selective LBBP with an iso-electrical window between the pacing spike and QRS onset;
     2. If using dual-lead method with one at His-bundle and the other at LBB region, a retrograde His-bundle potential is recorded from His-bundle lead during LBBP;
     3. LVATs at lead tip pacing of 1.5V/0.5ms and 10V/0.5ms are ≤ 80ms and the difference is < 10ms;
     4. A discrete LBB potential is recorded from lead tip and LVAT at tip pacing of 3V/0.5ms is ≤ 80ms19.
  If criterion 1 is fulfilled but none in criteria 2 is met, the procedure is considered to be left ventricular septal pacing (LVSP).
  Arms: LBBP group
Procedure: Right ventricular pacing — Implantation of a RV pacing lead is attempted using the standard-of-care technique first.
  Arms: RVP group

SUMMARY:
OptimPacing study has been designed as a prospective, multi-center, randomized, controlled trial. A total of 11 medical centers across China will enroll 683 patients over an estimated recruitment period of 2 years. An LBBP group will be compared with a group of conventional RVP in the follow-up of at least 3 years. The study aimed to demonstrate (1) the superiority of LBBP in preserving LV systolic function over RVP and (2) the feasibility and long-term safety of LBBP in patients with AV block.

DETAILED DESCRIPTION:
Introduction

Right ventricular pacing (RVP) has been the standard-of-care therapy for patients with bradycardia for sixty years. However, the selection of optimal pacing site is still controversial. Right ventricular septal or outflow tract pacing has not resulted in improved outcomes. RVP is considered to result in electrical and mechanical dyssynchrony and an increased risk of pacing-induced cardiomyopathy (PICM), heart failure and mortality. Biopace (Biventricular Pacing for Atrioventricular Block to Prevent Cardiac Desynchronization) study is a randomized controlled trial with a large population evaluating biventricular pacing versus RVP in patients with atrioventricular (AV) block. But biventricular pacing was not shown superiority in clinical outcomes compared with RVP. As biventricular pacing is delivered at two non-physiological sites, it actually creates ventricular dyssynchrony in patients with narrow QRS durations. Thus, seeking for the optimal pacing site has been the ultimate goal of doctors who specialize in cardiac pacing.

His-bundle pacing (HBP) is thought to be the most physiological pacing modality, which was initial applied by Deshmukh et al in 2000. HBP activates native His-Purkinje system and produces favorable electrical and mechanical synchrony. Clinical observations have shown HBP could reduce the incidence of PICM and improve combined clinical outcomes. However, HBP is not widely applied because of challenging operating techniques, unstable long-term pacing parameters and risk of loss of ventricular capture in a significant number of patients.

Left bundle branch pacing (LBBP) was first introduced by Huang et al in 2017. Since then, LBBP has been carried out boomingly in China. Similar with HBP, LBBP could activate left bundle branch (LBB) fibers and provide narrower paced QRS duration and better left ventricular (LV) mechanical synchrony than RVP. Animal studies also confirmed the physiological characteristics and anatomical lead locations of LBBP. Several clinical studies showed that LBBP could produce significantly narrower paced QRS duration and better echocardiographic response than biventricular pacing in patients with heart failure and LBB block. Furthermore, the implantation procedure appears easier and capture threshold is lower when compared with HBP. LBBP has appeared to be a promising approach in the clinical practice. However, no randomized controlled studies have been reported to compare the efficacy of LBBP and other pacing modalities.

Objectives

The study aimed to demonstrate (1) the superiority of LBBP in preserving LV systolic function over RVP and (2) the feasibility and long-term safety of LBBP in patients with AV block.

Methods

Stratified randomization

A balanced randomization is applied according to the following stratifying criteria:

1. AF with slow ventricular rate: present or absent;
2. LVEF: ≤ 50% or > 50%.

Lead implantation of LBBP

The lead implantation of LBBP has been well described previously. The implantation was performed using the Select Secure (3830) pacing lead delivered through a fixed-curve sheath. The 3830 lead was introduced transvenously into the right ventricle and screwed into the interventricular septum (IVS) until LV septum was reached, without protruding into the LV cavity.

Venous access was obtained via the left axillary vein or subclavian vein. The 3830 lead was inserted through the C315 HIS sheath. An intracardiac electrogram was recorded from the lead tip using the electrophysiological recording system. His-bundle electrogram was identified at the right anterior oblique 25° position and fluoroscopic image of the lead position was recorded as a reference. The sheath and lead tip were first advanced to the anterior lower site of the His-bundle position, and subsequently rotated in a counterclockwise fashion to place the lead tip in a perpendicular orientation to the IVS. A paced morphology of QS complex with a north in the nadir ("W"-shaped morphology) in surface lead V1 was usually observed at this location. As the lead tip was gradually screwed into the IVS, a rightward shift of the second notch in the "W"-shaped pacing morphology can be observed. The lead tip was considered to be in the final position once a paced morphology of right bundle branch delay (RBBD) in surface lead V1 was achieved. Moreover, a discrete potential before the QRS complex could be often recorded from the lead tip, and we defined this potential as the LBB potential. Left ventricular activation time (LVAT) was measured from the intracardiac pacing spike to the R-wave peak of QRS complex in lead V5 or V6. The penetration depth in the IVS was finally assessed by injecting a small amount of contrast medium through the sheath in left anterior oblique 45°. Echocardiography was routinely performed to evaluate the lead depth in the IVS before discharge.

Device programming

The devices are routinely programmed with a lower rate limit of 60 ppm. For DDD devices, the paced and sensed AV intervals are set as 150 and 120 ms, respectively.

Study organization

Echocardiographic core lab Echocardiographic examinations are performed at each study center before pacemaker implantation and at follow-up. All images are stored on DVD disks and sent to the core lab (Zhongshan Hospital, Fudan University) for central analysis.

Study Steering Committee

The study steering committee is composed of three experts who are not the investigators of this study. The committee is responsible for the academic issues including the judgment of LBBP or LVSP.

Independent Data Monitoring Committee (iDMC)

The iDMC is composed of three experts including at least one statistical expert. The committee is responsible for the data examination including mid-term evaluation during the study and also the patient privacy protection.

Safety Review Committee

The safety review committee is composed of three experts who are not the investigators of this study. In case of severe adverse events, including all-cause death, acute cardiovascular or cerebrovascular events and other lethal or disabling diseases, the committee will be responsible for the investigation of the events. The physicians should report the events to the principal investigator of each center and the committee within 2 hours. The committee should report the events to the hospital ethics committee in 24 hours. The committee may recommend the early termination of the study if an excessive rate of adverse events is suspected.

Statistical analysis

Intention-to-treat principle

Data analyses are performed according to the intention-to-treat principle. If LBBP or LVSP fails, RVP will be performed and the patient will not be crossed over to the other group. If LBBP fails but LVSP succeeds, the sub-group analysis for these patients with LVSP will be done.

Sample size

According to previous publications of HBP and RVP, we supposed that the rate of 5-year composite endpoints in RVP group was 25% and the rate in LBBP group was 15%. With a recruitment period of 2 years and follow-up time of at least 3 years, at least 100 events are required to achieve a power of 80%. With alpha as 0.05, rate of lost-of-follow-up rate as 10%, the final sample size was estimated as 683 by using PASS Version 15.

Endpoint analysis

Kaplan-Meier analysis was used to compare the rate of endpoints between the two groups over time. Cox proportional risk model will be applied to calculate the hazard ratio. A p-value less than 0.05 was considered statistically significant.

Mid-term analysis

Mid-term analysis is performed by iDMC when the rate of events reaches 50% (at least 50 events of primary endpoint). If LBBP group exhibits statistically significant superiority over RVP group with the significant level of 0.003, the study could be effectively early terminated. Otherwise, the sample size will be re-evaluated. The iDMC may determine if the study will continue according to the re-evaluation of the sample size. Eventually, the data prior to and after the mid-term analysis are put together for final analysis with the significant level of 0.047.

Statistical software

All statistical analyses were performed using SAS Version 9.4 or R Software Version 3.6.

Study timeframe

The study will start in October 2020 and the complete enrollment will be expected by the end of 2022. At least 11 medical centers across China will participate in the study. With a period of at least 3-year follow-up, the study is expected to finish at the end of 2025. The recruitment might be slower if the mid-term analysis does not reach the statistical significance and a larger population is required.

ELIGIBILITY:
Inclusion Criteria:

1. Indication of permanent pacemaker implantation: (1) Second degree or complete AV block; (2) Persistent or permanent atrial fibrillation with mean ventricular rate < 50 bpm and related symptoms
2. LVEF > 35%, NYHA classification I-III
3. Age > 18 years
4. Signed informed consent

Exclusion Criteria:

1. Implanted prosthetic tricuspid valve
2. Unstable angina, acute myocardial infarction, CABG or PCI within the last 3 months
3. Cardiac surgery like valvular replacement, TAVI, ventricular septal myectomy or ablation within the last 3 months
4. Enrolled in any other study
5. A life expectancy of less than 12 months or unable to undergo the planned 6. follow-up for any reasons
6. Pregnant or with a child-bearing plan
7. A history of heart transplantation
8. Complex congenital heart disease (whether surgical correction or not) and post-surgery repair or post-closure of ventricular septal defect
9. Ventricular septal hypertrophy (≥ 15mm during diastole)
10. Isolated persistent left superior vena cava
11. With ICD, CRT or CRTD indications
12. Pacemaker replacement, upgrade and pocket infection needing re-implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 683 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
A combined clinical endpoint of all-cause mortality, hospitalization for heart failure(HF) and/or occurrence of pacing-induced cardiomyopathy(PICM) | 6-month follow-up
  Incidence of all-cause death, hospitalization for HF and/or PICM
A combined clinical endpoint of all-cause mortality, hospitalization for heart failure(HF) and/or occurrence of pacing-induced cardiomyopathy(PICM) | 12-month follow-up
  Incidence of all-cause death, hospitalization for HF and/or PICM
A combined clinical endpoint of all-cause mortality, hospitalization for heart failure(HF) and/or occurrence of pacing-induced cardiomyopathy(PICM) | 24-month follow-up
  Incidence of all-cause death, hospitalization for HF and/or PICM
A combined clinical endpoint of all-cause mortality, hospitalization for heart failure(HF) and/or occurrence of pacing-induced cardiomyopathy(PICM) | 36-month follow-up
  Incidence of all-cause death, hospitalization for HF and/or PICM

SECONDARY OUTCOMES:
Left ventricular ejection fraction(LVEF) | Baseline; 6-month, 12-month, 24-month and 36-month follow-up
  Changes from baseline LVEF(unit: %) assessed by echocardiography at follow-up
Left ventricular end systolic volume(LVESV) | Baseline; 6-month, 12-month, 24-month and 36-month follow-up
  Changes from baseline LVESV(unit: mL) assessed by echocardiography at follow-up
Left ventricular end diastolic volume(LVEDV) | Baseline; 6-month, 12-month, 24-month and 36-month follow-up
  Changes from baseline LVEDV(unit: mL) assessed by echocardiography at follow-up
Left ventricular end systolic diameter(LVESD) | Baseline; 6-month, 12-month, 24-month and 36-month follow-up
  Changes from baseline LVESD(unit: mm) assessed by echocardiography at follow-up
Left ventricular end diastolic diameter(LVEDD) | Baseline; 6-month, 12-month, 24-month and 36-month follow-up
  Changes from baseline LVEDD(unit: mm) assessed by echocardiography at follow-up
Interventricular movement time difference(IVMD) | Baseline; 6-month, 12-month, 24-month and 36-month follow-up
  Changes from baseline IVMD(unit: ms) assessed by echocardiography at follow-up
Septal-to-posterior wall motion delay(SPWMD) | Baseline; 6-month, 12-month, 24-month and 36-month follow-up
  Changes from baseline SPWMD(unit: ms) assessed by echocardiography at follow-up
Changes in concentration of NT-proBNP in blood between baseline and follow-up | Baseline; 6-month,12-month, 24-month and 36-month follow-up
  Blood test is performed at each time frame to determine the concentration of NT-proBNP(unit: pg/mL)
Changes in New York Heart Association Heart Function Classification between baseline and follow-up | Baseline; 6-month,12-month, 24-month and 36-month follow-up
  The higher the classification, the more severe the heart failure symptoms(four levels: I, II, III and IV)
Changes in 6-minute Walk Distance between baseline and follow-up | Baseline; 6-month,12-month, 24-month and 36-month follow-up
  Distance that a participant walk within 6 minutes
Change in Quality Of Life Questionnaire score between baseline and follow-up | Baseline; 6-month,12-month, 24-month and 36-month follow-up
  Reflect the effect of cardiac funtion on quality of life, and higher scores represent a worse outcome
Pacing parameters | Before discharge; 1-month, 3-month, 6-month, 12-month, 24-month and 36-month follow-up
  Percentage of ventricular pacing, burden of atrial fibrillation, events of NSVT or VT
Incidence of other clinical adverse events | 6-month, 12-month, 24-month and 36-month follow-up
  New-onset atrial fibrillation, stroke, Upgrade to CRT, ICD, CRTD or HBP

CONTACTS AND LOCATIONS:
Overall Officials: Jiangang Zou, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sweeney MO, Hellkamp AS, Ellenbogen KA, Greenspon AJ, Freedman RA, Lee KL, Lamas GA; MOde Selection Trial Investigators. Adverse effect of ventricular pacing on heart failure and atrial fibrillation among patients with normal baseline QRS duration in a clinical trial of pacemaker therapy for sinus node dysfunction. Circulation. 2003 Jun 17;107(23):2932-7. doi: 10.1161/01.CIR.0000072769.17295.B1. Epub 2003 Jun 2. PMID 12782566
- [Background] Khurshid S, Epstein AE, Verdino RJ, Lin D, Goldberg LR, Marchlinski FE, Frankel DS. Incidence and predictors of right ventricular pacing-induced cardiomyopathy. Heart Rhythm. 2014 Sep;11(9):1619-25. doi: 10.1016/j.hrthm.2014.05.040. Epub 2014 Jun 2. PMID 24893122
- [Background] Funck RC, Blanc JJ, Mueller HH, Schade-Brittinger C, Bailleul C, Maisch B; BioPace Study Group. Biventricular stimulation to prevent cardiac desynchronization: rationale, design, and endpoints of the 'Biventricular Pacing for Atrioventricular Block to Prevent Cardiac Desynchronization (BioPace)' study. Europace. 2006 Aug;8(8):629-35. doi: 10.1093/europace/eul075. PMID 16864616
- [Background] Ruschitzka F, Abraham WT, Singh JP, Bax JJ, Borer JS, Brugada J, Dickstein K, Ford I, Gorcsan J 3rd, Gras D, Krum H, Sogaard P, Holzmeister J; EchoCRT Study Group. Cardiac-resynchronization therapy in heart failure with a narrow QRS complex. N Engl J Med. 2013 Oct 10;369(15):1395-405. doi: 10.1056/NEJMoa1306687. Epub 2013 Sep 2. PMID 23998714
- [Background] Deshmukh P, Casavant DA, Romanyshyn M, Anderson K. Permanent, direct His-bundle pacing: a novel approach to cardiac pacing in patients with normal His-Purkinje activation. Circulation. 2000 Feb 29;101(8):869-77. doi: 10.1161/01.cir.101.8.869. PMID 10694526
- [Background] Zhang J, Guo J, Hou X, Wang Y, Qian Z, Li K, Ge P, Zou J. Comparison of the effects of selective and non-selective His bundle pacing on cardiac electrical and mechanical synchrony. Europace. 2018 Jun 1;20(6):1010-1017. doi: 10.1093/europace/eux120. PMID 28575215
- [Background] Vijayaraman P, Naperkowski A, Subzposh FA, Abdelrahman M, Sharma PS, Oren JW, Dandamudi G, Ellenbogen KA. Permanent His-bundle pacing: Long-term lead performance and clinical outcomes. Heart Rhythm. 2018 May;15(5):696-702. doi: 10.1016/j.hrthm.2017.12.022. Epub 2017 Dec 20. PMID 29274474
- [Background] Abdelrahman M, Subzposh FA, Beer D, Durr B, Naperkowski A, Sun H, Oren JW, Dandamudi G, Vijayaraman P. Clinical Outcomes of His Bundle Pacing Compared to Right Ventricular Pacing. J Am Coll Cardiol. 2018 May 22;71(20):2319-2330. doi: 10.1016/j.jacc.2018.02.048. Epub 2018 Mar 10. PMID 29535066
- [Background] Sharma PS, Dandamudi G, Naperkowski A, Oren JW, Storm RH, Ellenbogen KA, Vijayaraman P. Permanent His-bundle pacing is feasible, safe, and superior to right ventricular pacing in routine clinical practice. Heart Rhythm. 2015 Feb;12(2):305-12. doi: 10.1016/j.hrthm.2014.10.021. Epub 2014 Oct 22. PMID 25446158
- [Background] Vijayaraman P, Chung MK, Dandamudi G, Upadhyay GA, Krishnan K, Crossley G, Bova Campbell K, Lee BK, Refaat MM, Saksena S, Fisher JD, Lakkireddy D; ACC's Electrophysiology Council. His Bundle Pacing. J Am Coll Cardiol. 2018 Aug 21;72(8):927-947. doi: 10.1016/j.jacc.2018.06.017. PMID 30115232
- [Background] Huang W, Su L, Wu S, Xu L, Xiao F, Zhou X, Ellenbogen KA. A Novel Pacing Strategy With Low and Stable Output: Pacing the Left Bundle Branch Immediately Beyond the Conduction Block. Can J Cardiol. 2017 Dec;33(12):1736.e1-1736.e3. doi: 10.1016/j.cjca.2017.09.013. Epub 2017 Sep 22. PMID 29173611
- [Background] Hou X, Qian Z, Wang Y, Qiu Y, Chen X, Jiang H, Jiang Z, Wu H, Zhao Z, Zhou W, Zou J. Feasibility and cardiac synchrony of permanent left bundle branch pacing through the interventricular septum. Europace. 2019 Nov 1;21(11):1694-1702. doi: 10.1093/europace/euz188. PMID 31322651
- [Background] Cai B, Huang X, Li L, Guo J, Chen S, Meng F, Wang H, Lin B, Su M. Evaluation of cardiac synchrony in left bundle branch pacing: Insights from echocardiographic research. J Cardiovasc Electrophysiol. 2020 Feb;31(2):560-569. doi: 10.1111/jce.14342. Epub 2020 Jan 20. PMID 31919928
- [Background] Qian Z, Hou X, Wang Y, Jiang H, Wu H, Chen X, Wang B, Zou J. Physiological Left Bundle Branch Pacing Validated by Ultra-High Density Ventricular Mapping in a Swine Model. Circ Arrhythm Electrophysiol. 2020 Jan;13(1):e007898. doi: 10.1161/CIRCEP.119.007898. Epub 2020 Jan 14. No abstract available. PMID 31935122
- [Background] Chen X, Jin Q, Li B, Jia J, Sharma PS, Huang W, Su Y, Ge J. Electrophysiological parameters and anatomical evaluation of left bundle branch pacing in an in vivo canine model. J Cardiovasc Electrophysiol. 2020 Jan;31(1):214-219. doi: 10.1111/jce.14300. Epub 2019 Dec 18. PMID 31778271
- [Background] Huang W, Wu S, Vijayaraman P, Su L, Chen X, Cai B, Zou J, Lan R, Fu G, Mao G, Ellenbogen KA, Whinnett ZI, Tung R. Cardiac Resynchronization Therapy in Patients With Nonischemic Cardiomyopathy Using Left Bundle Branch Pacing. JACC Clin Electrophysiol. 2020 Jul;6(7):849-858. doi: 10.1016/j.jacep.2020.04.011. PMID 32703568
- [Background] Wang Y, Gu K, Qian Z, Hou X, Chen X, Qiu Y, Jiang Z, Zhang X, Wu H, Chen M, Zou J. The efficacy of left bundle branch area pacing compared with biventricular pacing in patients with heart failure: A matched case-control study. J Cardiovasc Electrophysiol. 2020 Aug;31(8):2068-2077. doi: 10.1111/jce.14628. Epub 2020 Jul 6. PMID 32562442
- [Background] Li X, Qiu C, Xie R, Ma W, Wang Z, Li H, Wang H, Hua W, Zhang S, Yao Y, Fan X. Left bundle branch area pacing delivery of cardiac resynchronization therapy and comparison with biventricular pacing. ESC Heart Fail. 2020 Aug;7(4):1711-1722. doi: 10.1002/ehf2.12731. Epub 2020 May 13. PMID 32400967
- [Background] Ponnusamy SS, Arora V, Namboodiri N, Kumar V, Kapoor A, Vijayaraman P. Left bundle branch pacing: A comprehensive review. J Cardiovasc Electrophysiol. 2020 Sep;31(9):2462-2473. doi: 10.1111/jce.14681. Epub 2020 Jul 30. PMID 32681681